CLINICAL TRIAL: NCT01255345
Title: Female Chronic Pelvic Pain: Prevalence, Risk Factors and Clinical Characteristics With Particular Reference to the Pelvic Musculature
Brief Title: Female Chronic Pelvic Pain
Acronym: Female CPP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Copenhagen University Hospital at Herlev (Other)
Responsible Party: Sys Loving, PT, MSc, ph.d.-student, Multidisciplinary Pain Center, Herlev Hospital
Other Study IDs: H-1-2010-037
Record Dates: First submitted 2010-12-06; First posted 2010-12-07 (Estimated); Last update posted 2011-06-27 (Estimated); Status verified 2010-10

CONDITIONS: Pelvic Pain; Abdominal Pain; Painful Bladder Syndrome; Interstitial Cystitis; Irritable Bowel Syndrome
Keywords: Physiotherapy; Multidisciplinary Pain Centers; Pain measurements; Physical activity; Quality of life
MeSH Terms: conditions — Pelvic Pain; Abdominal Pain; Cystitis, Interstitial; Irritable Bowel Syndrome; Motor Activity

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (1):
- Adult females with CPP living in Denmark
  Interventions: Other: Chronic pelvic pain

INTERVENTIONS:
Other: Chronic pelvic pain — A physioterapeutic examination of abnormal muscular findings, i.e tonus, elasticitt and strength, in the pelvic area connected to female CPP.

SUMMARY:
The purpose of this study is to investigate the frequency and severity of chronic pelvic pain (CPP) in adult women living in Copenhagen Country and Zealand Country (total population 2,4 million), Denmark, in relation to selected factors, such as basic demographic and clinical factors, health related quality of life, physical activity and abnormal muscular findings in the pelvic area.

DETAILED DESCRIPTION:
Introduction:

The aim of this study is to investigate the frequency and severity of chronic pelvic pain (CPP) in adult women living in Copenhagen Country and Zealand Country (total population 2,4 million), Denmark, in relation to selected factors, such as basic demographic and clinical factors, health related quality of life, physical activity and abnormal muscular findings in the pelvic area.

Methods:

The study is designed as a cross-sectional, questionnaire-based survey and two randomly selected age stratified groups of the responding participating women, one with or one without pain, will receive a clinical examination by a specialist physiotherapist for abnormal muscular finding in the pelvic, lower abdominal or inguinal area.

Results:

Descriptive characteristics will be obtained by univariate analysis and presented as means with standard deviations, or percentages. T test and the Mann-Whitney test will be used to analyze continuous data with and without normal distribution, respectively, and the Chi-square test or Fisher's exact test will be used to analyze categorical data, as appropriate. Correlation between self-reported CPP and abnormal muscular findings will be analysed. Logistic regression analysis will be used to identify the independent variables significantly associated with CPP. For logistic regression analysis, we will select only those findings that are significant as determined by Fisher's exact or the Chi-square test, with values of 0 and 1 assigned to the absence and presence, respectively, of each variable in each subject.

ELIGIBILITY:
Inclusion Criteria:

* Women ≥ 18 years
* Living in Copenhagen Country (Region H)
* Capable of reading, writing and speaking Danish

Exclusion Criteria:

* Pain limited solely to the perineal skin or introitus (vulvodynia)
* Pregnancy, cancer, active pelvic inflammatory disease
* Operation in the pelvic during the last 6 months
* Cognitively impaired individuals

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: 2500 adult women living in Copenhagen Country and Zealand Country (total population 2,4 million), Denmark
Sampling Method: Probability Sample
Enrollment: 2500 (Estimated)
Dates: Start 2011-01; Study Completion 2012-12 (Estimated)

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Anaesthesiology, Herlev University Hospital, Herlev, Copenhagen, Denmark